CLINICAL TRIAL: NCT04678765
Title: Efficacy of Ultrasound-guided Axillary Nerve Block Versus Ultrasound-guided Peripheral Forearm Block in Patients Undergoing Hand Surgery: A Randomized Controlled Trial
Brief Title: Efficacy of Ultrasound-guided Axillary Nerve Block Versus Ultrasound-guided Peripheral Forearm Block in Patients Undergoing Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JessaH_Axillaryblock
Record Dates: First submitted 2020-11-30; First posted 2020-12-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Surgery; Anesthesia, Local

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided distal peripheral nerve block (Active Comparator): Patients will receive the ultrasound-guided distal peripheral nerve block (locoregional anesthesia)
  Interventions: Procedure: Ultrasound-guided distal peripheral nerve block
- Ultrasound-guided quadruple-injection axillary nerve block (Experimental): Patients will receive the ultrasound-guided quadruple-injection axillary nerve block (locoregional anesthesia)
  Interventions: Procedure: Ultrasound-guided quadruple-injection axillary nerve block

INTERVENTIONS:
Procedure: Ultrasound-guided distal peripheral nerve block — To localize the median nerve, the ultrasound transducer will be placed in a transverse orientation proximally to the wrist cease at mid-forearm level, with a slight tilt distally towards the hand. An in-plane ultrasound-guided medial-to-lateral puncture will be made and 3ml of 2% lidocaine was injected within the fascia that envelopes the median nerve.
  To perform the ulnar block, an ultrasound transducer will be placed in a transverse orientation over the ulnar side of the distal forearm. An in-plane ultrasound-guided medial-to-lateral or proximal-to distal puncture will be made and 3 ml of 2% lidocaine will be infiltrated into the fascial plane to block the ulnar nerve. Finally, we will apply a circumferential subcutaneous infiltration of 4 ml 2% lidocaine at the radial side of the wrist, 2cm proximal to the styloid process of the radius to block the terminal sensory branches of the radial, musculocutaneous, and medial antebrachial cutaneous nerves that may reach the palmar crease.
  Arms: Ultrasound-guided distal peripheral nerve block
Procedure: Ultrasound-guided quadruple-injection axillary nerve block — The US probe will be applied in the axilla to obtain a short-axis view of the axillary artery. The following 4 nerves will be identified as hyperechoic structures: the median, ulnar, and radial nerve surrounding the axillary artery and the musculocutaneous nerve in the fascial layers between the biceps and coracobrachialis muscles.
  A total volume of 20 mL lidocaine 2% will be administered divided over 4 locations. The needle is inserted in-plane from the anterior aspect of the axillary artery and directed toward the posterior aspect of the axillary artery to first anesthetize the radial nerve. The posteriorly located radial nerve is surrounded with 8 mL of local anesthetic. Afterward, the needle is withdrawn and redirected to the median and ulnar nerves, after which another 8 mL of local anesthetic is deposited. In the end, the needle is withdrawn and redirected toward the musculocutaneous nerve where another 4 mL of local anesthetic is deposited.
  Arms: Ultrasound-guided quadruple-injection axillary nerve block

SUMMARY:
By means of an observer-blinded, mono-center, prospective, randomized controlled superiority trial, the total anesthesia-related time (sum of performance and onset times) of an ultrasound-guided distal peripheral nerve block and an ultrasound-guided axillary nerve block will be investigated in patients undergoing hand surgery. The hypothesis is that the onset-time of the ultrasound-guided distal peripheral nerve block will be faster than ultrasound-guided axillary nerve blocks, which is more suitable for hand surgery.

DETAILED DESCRIPTION:
Introduction:

Regional anesthesia (RA) has become an increasingly popular alternative for general anesthesia in day-care hand surgery. It has been demonstrated to allow faster recovery and to reduce time to discharge from the hospital (lower pain scores, less nausea, … ), resulting in lower hospital costs.

An ultrasound-guided distal peripheral nerve block of the n. medianus and n. ulnaris is frequently used in locoregional anesthetic technique in superficial hand surgery. Distal peripheral nerve blocks allow preservation of proximal muscle function of the upper limb, which may also allow patients to move affected digits when instructed to do so during surgery.

Another frequently used locoregional technique in superficial hand surgery is the axillary nerve block. An ultrasound-guided axillary nerve block anesthetizes the n. medianus, n. ulnaris, n. radialis, and n. musculocutaneous at an early stage in their trajectory in the arm, providing satisfactory anesthesia for elbow, forearm, and hand surgery and provides reliable cutaneous anesthesia of the inner upper arm including the medial cutaneous nerve of the arm and intercostobrachial nerve, areas often missed with other approaches.

Ambulatory superficial hand surgery is frequently conducted in JESSA hospital and is most frequently conducted using intravenous regional anesthesia (IVRA) of the forearm, an ultrasound-guided distal peripheral nerve block, or an ultrasound-guided axillary nerve block.

Traditionally, these locoregional anesthesia techniques have been studied and compared with respect to analgesic efficacy and safety. Block performance time and onset-time of sensory block after locoregional anesthesia for hand-surgery is important in operating room turn-over and efficiency. Also, patient satisfaction, which can be influenced by multiple factors and not only by the chosen anesthetic technique, is important to evaluate. Even the inability to use the affected limb due to the motor block of proximal and distal musculature has been shown to reduce patient satisfaction.

Outcome measures:

The primary endpoint of this study is comparing the total anesthesia-related time (sum of block performance time and onset time) of an ultrasound-guided distal peripheral nerve block and an ultrasound-guided axillary nerve block. Block performance time is defined as the time interval between the start of the block procedure and the end of the block procedure, thus imaging + needling time.

Block performance time will be recorded with a stopwatch by the attending block room nurse. Time for the sensory block to take effect is defined as the time required for the limb to achieve a level of anesthesia deemed adequate for surgery (i.e., not necessarily a complete block) after placement of the block.

After placement of the block, a single, blinded study nurse will enter the block room and will carry out measurements of plexus blockade every 2 mins until 30 mins. Sensory blockade of the median and ulnar nerves will be graded according to a 3-point scale using a cold test: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch). Sensory blockade of the median and ulnar nerves will be assessed on the volar aspect of the thumb, and the volar aspect of the fifth finger, respectively. We consider the patient ready for surgery when a minimal sensory block score of 3 out of 4 points is achieved, provided the sensory block score is equal or superior to 3 out of 4 points.

Secondary endpoint:

* Surgical block success rate: (sensory) Block success, defined as the ability of the surgeon to perform surgery without the use of any rescue block or supplemental general anesthesia, evaluated at the end of surgery. 3 scores are available: 1. Complete sensory block, 2. Incomplete block with IV rescue medication or extra local anesthetic and 3. Unsuccessful block with need for general anesthesia.
* Patient satisfaction: Patient satisfaction was evaluated using the "Evaluation du Vécu de l' Anesthésie LocoRegional" (EVAN-LR) questionnaire which was specially developed for the evaluation of patient satisfaction after RA.
* Different time intervals will be measured: needling time (defined as the time from injection of the needle to the removal of the needle), surgical time (defined as the time from incision to surgical completion and application of dressings), total OR stay time (defined as departure time from the OR minus arrival time in the OR), and tourniquet time (defined as the total time the tourniquet is inflated).
* Intraoperative need for supplemental analgesia
* The conversion rate to general analgesia (i.e., block failure rate)
* Patient's pre-, intra-, and postoperative pain scores at several time points, measured via an 11-point Numeric Rating Scale (NRS) in which number 0 means "no pain at all", number 5 means "moderate pain", and number 10 means "worst possible pain".
* Tourniquet tolerance time (defined as the time required for the tourniquet pressure to become painful (NRS > 3)
* Required doses of analgesics were measured (paracetamol, ibuprofen, tramadol).
* Surgical satisfaction, using a "seven-point Likert scale" (on a scale from 1 to 7, 1 on 7 is absolutely not satisfied, 4 on 7 neutral, and 7 on 7 being very satisfied) on surgical conditions after surgery.
* Adverse events

Design:

In this observer-blinded, mono-center, prospective, randomized controlled superiority trial 2 anesthetic procedures will be compared in patients that undergo hand surgery (carpal tunnel release, finger amputation, finger manipulation, hand foreign body removal, hand incision and drainage, metacarpal fracture repair, trigger finger release, tendon repair, and Dupuytren's contracture).

This study will be performed according to the Declaration of Helsinki and will be approved by the ethics committee of the JESSA Hospital, Hasselt, Belgium before the start of the study. Written informed consent will be obtained before participation in the study.

Randomization will be performed using a computer-generated random allocation sequence. Allocation numbers will be sealed in opaque envelopes, which will be opened in sequence by an independent anesthesiologist who is not involved in the assessment of outcomes.

The surgeon and the researcher will be blinded for the used type of anesthesia. To achieve observer blinding, surgeons and study nurses are not allowed in the regional anesthesia block room and are asked to leave the operation theatre at the end of each procedure.

Study procedures:

The patient will first receive information about this study. Before the start of the study, written informed consent will be obtained, after which the patient will be randomized to one of the 2 treatment groups. All patients will receive an intravenous catheter in the contralateral arm with IV. Infusion of NaCl 0.9% 500ml 60ml/h, supplementary oxygen, and standard monitoring (non-invasive blood pressure, electrocardiogram, and saturation measurements).

Ultrasound-guided distal peripheral nerve block:

Both ultrasound, pressure-monitoring, and neuro-stimulation (set at 0.5 mA) will be used to detect the nerves and to avoid intra-neural puncture/injection. A Sono Site Xporte ultrasound machine with a high-frequency linear transducer HFL38 (13-6MHz) and a 22G Stimuplex Ultra 50 mm (B. Braun Medical Inc, Melsungen, Germany) needle will be used to locate the median nerve and ulnar nerve. An in-plane ultrasound-guided medial-to-lateral puncture will be made and 3ml of 2% lidocaine will be injected within the fascia that envelopes the median nerve. In addition, depending on the available space, an in-plane ultrasound-guided medial-to-lateral or proximal-to distal puncture will be made and 3 ml of 2% lidocaine will be infiltrated into the fascial plane to block the ulnar nerve.

Ultrasound-guided quadruple-injection axillary nerve block:

A Sono Site Xporte ultrasound machine with a high-frequency linear transducer HFL38 (13-6MHz) and a 22G Stimuplex Ultra 50 mm (B. Braun Medical Inc, Melsungen, Germany) needle will be used. The US probe will be applied in a sterile fashion in the axilla to obtain a short-axis view of the axillary artery. The following 4 nerves will be identified as hyperechoic structures: the median, ulnar, and radial nerve surrounding the axillary artery and the musculocutaneous nerve in the fascial layers between the biceps and coracobrachialis muscles. The needle is inserted in-plane from the anterior aspect of the axillary nerve and directed toward the posterior aspect. Both ultrasound, pressure-monitoring, and neuro-stimulation (set at 0.5 mA) will be used to detect the nerves and to avoid intra-neural puncture/injection. A total volume of 20 mL lidocaine 2 % will be administered divided over four locations. The needle is inserted in plane from the anterior aspect of the axillary artery and directed toward the posterior aspect of the axillary artery to first anesthetize the radial nerve. The posteriorly located radial nerve is surrounded with 8 mL of local anesthetic. Afterward, the needle is withdrawn and redirected to the median and ulnar nerves, after which another 8 mL of local anesthetic is deposited. In the end, the needle is withdrawn and redirected toward the musculocutaneous nerve where another 4 mL of local anesthetic is deposited.

Before the start of the surgery, the single tourniquet, 5cm in width, will be placed 5 cm distal to the medial epicondyle of the humerus. A band-aid was already placed on the dorsal side of the ipsilateral hand of patients enrolled in the peripheral nerve block group at the regional anesthesia block room. If the block is insufficient [numeric rating scale (NRS) > 4], patients will receive an injection of supplemental local anesthetic at the operation site or an IV. bolus of 5μg sufentanil repeated once if necessary. If pain is persistent or the block failed, general anesthesia will be induced with 2 mg/kg propofol. A laryngeal mask will be inserted and anesthesia will be maintained with sevoflurane 1.5 to 2.0% in a 40% O2/air mixture.

Furthermore, peroperatively patients will receive intravenous paracetamol 15mg/kg (max 1gram), ketorolac 0.5mg/kg (max 30mg), and dexamethasone 0.1mg/kg (max 5mg) if no contraindications are present.

In case of conversion to general anesthesia or adverse events (hypotension, bradycardia, or symptoms of LAST), patients will be monitored in the post-anesthesia care unit (PACU) until the problem has resolved, otherwise, they are admitted directly postoperative to the day care unit (DCU). At the PACU, postoperative pain (NRS > 3) is treated with tramadol 50-100 mg PO. Postoperative nausea or vomiting (PONV) is treated with ondansetron 4 mg IV. After hospital discharge, patients' oral medication scheme consists of paracetamol (500mg for < 60kg and 1gram for > 60kg) 1x/6u and ibuprofen (400mg for < 60kg and 600mg for > 60kg LG and good kidney functioning) 1x/8u if needed for a maximum of 5 days.

Statistical analysis:

The necessary sample size was determined for the primary outcome, the anesthesia-related time, with the aim to demonstrate the superiority of an ultrasound-guided distal peripheral nerve block compared to an ultrasound-guided axillary nerve block. A 20% time difference between groups is considered statistically significant. According to a previous trial, the anesthesia-related time of the 4-injection ultrasound-guided axillary nerve block technique is 25.5 +/- 7.7 min. Assuming α=0.05 and power=0.80 for a 20% time difference in the anesthesia-related time using a two-sided Chi-Square test, the calculated sample size is 74. To account for a possible 10% drop-out rate, the sample size was increased to 40 patients per group, so 80 patients in total.

All statistical analyses will be performed with SPSS 25.0 (IBM® SPSS® Inc, Chicago, Illinois, USA). Continuous variables will be summarized by their mean and standard deviation, or median and interquartile range if severe deviations from normality would be observed. Comparisons between randomized groups will be made using a Student t-Test, or Wilcoxon rank-sum test in case of non-normality. Categorical data will be collected by observed frequencies and percentages per category. Comparisons between randomized groups were made using a chi-square test or Fisher's exact test, as appropriate. Continuous repeated data were corrected for multiple testing. A p-value <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* ASA (American Society of Anesthesiology) classification: 1 - 3
* Scheduled for surgery in the day surgery unit
* Patients planned for unilateral hand surgery: carpal tunnel release, finger amputation (except digit I and II), finger manipulation (except digit I and II), hand foreign body removal (except digit I and II), hand incision and drainage, metacarpal fracture repair (except digit I and II), trigger finger release (except digit I), tendon repair (except digit I), and Dupuytren's contracture (except digit I)

Exclusion Criteria:

* Refusal of the patient
* Bilateral surgery
* BMI ≥ 40 kg/m²
* Puncture site infections
* Preexisting peripheral neuropathy
* Chronic pain syndrome
* Diabetes mellitus
* Pregnancy
* Use of strong pain medication in the past 3 months
* Allergy for any of the medications used
* Coagulation disorders or the use of anticoagulant therapy (vitamin K antagonists, new oral anticoagulants) or antiplatelet drugs (thienopyridines)
* Contra-indication for the use of a tourniquet
* Previous surgery in the same upper extremity
* Impossibility to understand the study protocol
* Not understanding the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Total anaesthesia-related time | Preoperative
  The total anesthesia-related time is the sum of block performance time and onset time of the block. Block performance time is defined as the time interval between the start of the block procedure and the end of the block procedure, thus imaging + needling time. Block performance time will be recorded with a stopwatch by the attending block room nurse.
  Time for the sensory block to take effect is defined as the time required for the limb to achieve a level of anesthesia deemed adequate for surgery (i.e., not necessarily a complete block) after placement of the block.

SECONDARY OUTCOMES:
Surgical block success rate | Intraoperative
  (Sensory) block success, defined as the ability of the surgeon to perform surgery without the use of any rescue block or supplemental general anesthesia, evaluated at the end of surgery. 3 scores are available: 1 complete sensory block, 2. Incomplete block with IV rescue medication or extra local anesthetic and 3. Unsuccessful block with need for general anesthesia.
Patient satisfaction | Day 0 and day 1 postoperatively
  Patient satisfaction was evaluated using the "Evaluation du Vécu de l' Anesthésie LocoRegional" (EVAN-LR) questionnaire which was specially developed for the evaluation of patient satisfaction after RA. All questions were completed just before discharge, except for those regarding items, which are home-related (question 12-13-14). These questions will be asked during a postoperative phone call on day 1.
Needling time | Preoperative
  The time from injection of the needle to the removal of the needle.
Surgical time | Intraoperative
  The time from incision to surgical completion and application of dressings.
Total OR stay time | Intraoperative
  Departure time from the OR minus arrival time in the OR.
Tourniquet time | From start of inflation until deflation of the tourniquet
  Total time the tourniquet is inflated
Intraoperative need for supplemental analgesia | Intraoperative
  The need for supplemental analgesia during the surgery.
The conversion rate to general analgesia | Intraoperative
  Block failure rate
Pain due to anesthesia technique: Numeric Rating Scale (NRS) | At the end of performing the anesthesia technique
  Pain caused by performing the anesthesia technique (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Pain score at start of surgery (surgical incision): Numeric Rating Scale (NRS) | At the start of the surgical procedure
  Pain score at surgical incision (start of surgical procedure) (11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Intraoperative pain score: Numeric Rating Scale (NRS) | Every 5 minutes during the surgical procedure, until the end of surgery (last stitch) (up to 25 minutes)
  Pain score (11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable) at every 5 min during the surgical procedure (both surgical pain and tourniquet pain)
Postoperative pain score: Numeric Rating Scale (NRS) | Day 0 and day 1 postoperatively
  Pain score (11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable) at discharge and 24 hours after the surgery
Tourniquet tolerance time | From start of inflation until deflation of the tourniquet
  The time required for the tourniquet pressure to become painful (NRS >3)
Required doses of intraoperative pain medication | Intraoperative
  Total doses of analgesics required during surgery (paracetamol, ibuprofen, tramadol)
Required doses of postoperative pain medication | Day 0 postoperatively
  Total doses of analgesics required after surgery (paracetamol, ibuprofen, tramadol)
Required doses of postoperative pain medication | Day 1 postoperatively
  Total doses of analgesics required 24 hours after surgery (paracetamol, ibuprofen, tramadol)
Surgical satisfaction | At the end of the surgery
  Surgical satisfaction, using an "seven-point Likert scale" (on a scale from 1 to 7, 1 on 7 is absolutely not satisfied, 4 on 7 neutral and 7 on 7 being very satisfied) on surgical conditions after surgery.
Adverse events | Day 1 postoperative
  The incidences of hypotension, bradycardia, PONV, symptoms of local anesthetic toxicity (LAST) and neurological damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No